CLINICAL TRIAL: NCT00272532
Title: The Efficacy of Topical Thiocolchicoside in Cervical Myofascial Pain Syndrome: Triple-Arm, Single-Blind, Randomized, Prospective, Phase IV Clinical Study
Brief Title: EMINEM: Efficacy of Muscoril In NEck Myofascial Syndromes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: L_9892
Record Dates: First submitted 2006-01-04; First posted 2006-01-06 (Estimated); Last update posted 2008-02-20 (Estimated); Status verified 2008-02

CONDITIONS: Myofascial Pain Syndromes
MeSH Terms: conditions — Myofascial Pain Syndromes | interventions — thiocolchicoside

INTERVENTIONS:
Drug: Thiocolchicoside

SUMMARY:
Study objective:

* To demonstrate, in patients with myofascial pain syndrome in cervical region, the degree of efficacy of thiocolchicoside ointment administered to trigger point regions compared with the trigger point injection.

ELIGIBILITY:
Inclusion Criteria:

* Submitted to clinic with a complaint of head and neck pain
* Be diagnosed as having myofascial pain syndrome by determining the active trigger points in trapezius and/or interscapular region according to criteria of Simons and Travel
* Have 1 to 8 active trigger point(s)

Exclusion Criteria:

* Have evident cervical discopathy and signs of osteoarthritis
* Have bleeding diathesis or using anticoagulant medication which hinders injection
* Have known malignity, being used steroids, have immunodepressive disorders and/or being taken immunodepressive drugs
* Be pregnant or have the possibility of being pregnant or not being used a regular contraceptive method
* Have known allergic reaction against Thiocolchicoside

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 65
Dates: Start 2005-04

PRIMARY OUTCOMES:
Pain relief (Visual Analog Scale and sensitometer) and increase in mobility of neck. Patient and physician satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Edibe Taylan, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Istanbul, Turkey (Türkiye)